CLINICAL TRIAL: NCT00004807
Title: Study of the Pathogenesis of Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12009; JHUSM-KKI-87021203
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Rett Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Dextromethorphan; Topiramate; Donepezil

INTERVENTIONS:
Drug: dextromethorphan
Drug: topiramate
Drug: Donepezil

SUMMARY:
OBJECTIVES: I. Extend current knowledge of the phenotype and natural history of Rett syndrome (RS).

II. Continue the search for a cytogenetic and/or DNA marker. III. Study the effects of cholinergic drugs based on preliminary evidence for reduced levels of brain acetylcholine, while continuing supportive care to modify seizures, respiratory abnormalities, and motor disturbances, and improve nutrition, behavior, and learning.

IV. Identify targets for future therapeutic interventions, e.g., growth factors, to influence neurologic recovery.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive a comprehensive clinical evaluation including an ophthalmologic exam; speech, communication, and developmental assessment; nutritional evaluation; neurologic exam; respiratory monitoring; and cytogenetic studies.

Selected patients with malnutrition are given night feedings of Pediasure with Fiber by nasogastric tube. Specific recommendations for feeding techniques and diet are made.

Selected patients with seizures or severe hyperventilation and progressive rigidity are nonrandomly assigned to dextromethorphan or topiramate therapy.

Oral dextromethorphan is maintained 6 months to 1 year; duration of therapy depends on response. Oral topiramate is given for 6 months to 1 year, and Aricept for 6 months to 1 year.

Concurrent anticonvulsants may require dose adjustments while on above protocols. Supportive care for constipation, scoliosis, and weight loss is allowed.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Rett syndrome

Diagnosis confirmed on study

Ages: 0 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Sakkubai Naidu, Study Chair — Johns Hopkins University

REFERENCES:
- [Background] Wenk GL, Naidu S, Casanova MF, Kitt CA, Moser H. Altered neurochemical markers in Rett's syndrome. Neurology. 1991 Nov;41(11):1753-6. doi: 10.1212/wnl.41.11.1753. PMID 1658685
- [Background] Reiss AL, Faruque F, Naidu S, Abrams M, Beaty T, Bryan RN, Moser H. Neuroanatomy of Rett syndrome: a volumetric imaging study. Ann Neurol. 1993 Aug;34(2):227-34. doi: 10.1002/ana.410340220. PMID 8338347
- [Background] Wenk GL, O'Leary M, Nemeroff CB, Bissette G, Moser H, Naidu S. Neurochemical alterations in Rett syndrome. Brain Res Dev Brain Res. 1993 Jul 16;74(1):67-72. doi: 10.1016/0165-3806(93)90084-n. PMID 8403377
- [Background] Cooke DW, Naidu S, Plotnick L, Berkovitz GD. Abnormalities of thyroid function and glucose control in subjects with Rett syndrome. Horm Res. 1995;43(6):273-8. doi: 10.1159/000184309. PMID 7607612
- [Background] Naidu S, Hyman S, Harris EL, Narayanan V, Johns D, Castora F. Rett syndrome studies of natural history and search for a genetic marker. Neuropediatrics. 1995 Apr;26(2):63-6. doi: 10.1055/s-2007-979724. PMID 7566454
- [Background] Naidu S, Hyman S, Piazza K, Savedra J, Perman J, Wenk G, Kitt C, Troncoso J, Price D, Cassanova M, et al. The Rett syndrome: progress report on studies at the Kennedy Institute. Brain Dev. 1990;12(1):5-7. doi: 10.1016/s0387-7604(12)80164-1. PMID 2344026
- [Background] Casanova MF, Naidu S, Goldberg TE, Moser HW, Khoromi S, Kumar A, Kleinman JE, Weinberger DR. Quantitative magnetic resonance imaging in Rett syndrome. J Neuropsychiatry Clin Neurosci. 1991 Winter;3(1):66-72. doi: 10.1176/jnp.3.1.66. PMID 7580176
- [Background] Naidu S, Wong DF, Kitt C, Wenk G, Moser HW. Positron emission tomography in the Rett syndrome: clinical, biochemical and pathological correlates. Brain Dev. 1992 May;14 Suppl:S75-9. PMID 1385677
- [Background] Marcus CL, Carroll JL, McColley SA, Loughlin GM, Curtis S, Pyzik P, Naidu S. Polysomnographic characteristics of patients with Rett syndrome. J Pediatr. 1994 Aug;125(2):218-24. doi: 10.1016/s0022-3476(94)70196-2. PMID 8040765